CLINICAL TRIAL: NCT03677856
Title: A Randomised Controlled Trial to Investigate the Effectiveness of ThOracic Epidural and Paravertebral Blockade In Reducing Chronic Post- Thoracotomy Pain: 2
Brief Title: The Effectiveness of ThOracic Epidural and Paravertebral Blockade In Reducing Chronic Post- Thoracotomy Pain: 2
Acronym: TOPIC-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_18-0108
Record Dates: First submitted 2018-09-13; First posted 2018-09-19 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Anesthesia; Thoracic Diseases
Keywords: Paravertebral block; Thoracic epidural block; Thoracotomy
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Intervention Model Description: Multi-centre, parallel group, superiority, with an internal pilot, in a 1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral Blockade (Experimental): Anaesthesia to single side of the patient's chest
  Interventions: Procedure: Paravertebral blockade
- Thoracic epidural block (Active Comparator): Anaesthesia to both sides of the patient's chest
  Interventions: Procedure: Thoracic epidural block

INTERVENTIONS:
Procedure: Paravertebral blockade — Type of anaesthesia
  Arms: Paravertebral Blockade
Procedure: Thoracic epidural block — Type of anaesthesia
  Arms: Thoracic epidural block

SUMMARY:
An estimated 7200 thoracotomies (surgical incision into the chest wall) are performed annually in the UK, most commonly to treat lung cancer. It is considered one of the most painful surgical procedures due to tissue, muscle and nerve damage from the incision, and as the wound heals. The normal breathing motion and nerve injury caused during surgery can result in a high risk of persistent pain for months after surgery. Chronic post-thoracotomy pain (CPTP) is defined as pain that recurs or persists at least two months following the surgery and can occur in up to half of these patients.

There are two commonly used for pain control during thoracotomy: Thoracic Epidural Block (TEB) blocks nerves on both sides of the chest at the spinal cord. It reduces painful nerve signals but may not abolish them completely. Para Vertebral Blockade is done only on the side of surgery and may completely block painful nerve signals from reaching the spinal cord. This total blockade of nerve signals could decrease the likelihood of developing chronic pain and could be uniquely effective in preventing long-term pain.

Over a period of 30 months this trial will be attempting to approach all patients undergoing a thoracotomy at approximately 20 UK hospitals to see if they wish to participate, and to look at the reasons they may not want to participate. We will follow up each participant for a maximum of a year following their surgery.

There is a qualitative intervention embedded within this study to support recruitment.

DETAILED DESCRIPTION:
At the present time, both thoracic epidural block (TEB) and paravertebral blockade (PVB) are routinely used in the UK to provide pain relief for patients undergoing elective open thoracotomy. TEB has long been regarded as the 'gold standard' technique of pain relief for thoracotomy but this has recently been challenged from an overview of the literature on trends and new evidence in the management of acute and chronic post-thoracotomy pain.

In TOPIC 2 the interventional arm will be peri-operative (at or around the time of surgery) pain relief using PVB and the comparator arm will be peri-operative pain relief using TEB. The only pre-operative change to the patient pathway in TOPIC 2 is that the patient will be approached during pre-operative assessment at least 24 hours prior to surgery.

Post-operatively patients will receive analgesia in line with current practice. The trial's hypothesis is that in adult patients undergoing elective open thoracotomy, the use of paravertebral blockade for pain relief at or around the time of surgery reduces both the number of people reporting chronic pain and the persistence of chronic pain at six months by at least 10%, compared with the use of thoracic epidural block. To detect this difference a total of 1026 patients will be recruited from approximately 20 UK hospitals.

Interim analyses of safety and efficacy for presentation to the independent DMC will take place during the study. The committee will meet prior to study commencement to agree the manner and timing of such analyses but this is likely to include the analysis of the primary and major secondary outcomes and full assessment of safety (SAEs) at least at annual intervals. Criteria for stopping or modifying the study based on this information will be ratified by the DMC, but there is also an embedded pilot phase which sets out criteria for assessing whether sufficient progress is made during the first 12 months of recruitment. Failure to open enough sites to recruitment or recruit enough patients from those sites, may be sufficient reason to terminate the trial, or at least re-design some of it to ease these problems.

A randomised controlled trial design has been chosen since this is the acknowledged "gold standard" for evidence based medicine and, because only the patients themselves can say how much pain they are in, patient reported outcomes are appropriate in answering the trial question. Because of the nature of the procedure it is not possible to conceal the surgical team performing the procedure from the allocation but they will not know in advance which of the allocated treatments will be received. There is no reason to believe that patients will have any preconceptions regarding the levels of chronic pain they will experience so the chance of bias is low in this regard.

TOPIC 2 has been designed as a pragmatic trial which collates data during the hospital admission for thoracotomy then, by telephone interview and postal questionnaire at 3, 6 and 12 months. This schedule of events as well as both the type and amount of data collected has been created with substantial input from 2 patient/public representatives.

Since the track record of recruitment to trials involving surgery is not as good as in other areas of medicine, the trial has embedded a qualitative component which will specifically look at the consent process and the reasons for patients either entering or not entering the trial. Patients will therefore initially be asked to consent to the conversation introducing the trial being recorded, and to participate in the main trial. They can choose to participate in just the interview process (conducted in the clinic), just the main trial, neither, or both.

The trial documentation has been prepared in advance of submission to ethics and recruitment is estimated to start in the final quarter of 2018, for 30 months. The first 12 months of recruitment will form an internal pilot phase during which the feasibility of the overall trial will be assessed. Although the primary outcome requires only 6 months followup, patients will be followed up for year to provide a further estimate of how long any differences in pain levels lasts. It will take approximately a further 6 months to analyse the data prior to publication.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Elective open thoracotomy
* Able to provide written informed consent
* Willingness to complete study questionnaires up until 12 months post randomisation

Exclusion Criteria:

* Contraindication to TEB or PVB e.g. known allergy to local anaesthetics; infection near the proposed puncture site; coagulation disorders, thoracic spine disorders
* Surgery for chest wall pathology on the side of surgery
* Previous thoracotomy
* Median sternotomy within 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1026 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2022-01-08 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic pain: incidence = score > 40 on visual analogue score | 6 months post trial thoracotomy
  Patient reported pain lasting at least 3 months as measured by visual analogue score

SECONDARY OUTCOMES:
Complications of regional anaesthesia | 3, 6 and 12 months post randomisation
  Complications of regional anaesthesia are protocol-defined
Incidence of surgical complications | Until discharge from hospital post randomisation eg a maximum of 30 days
  as classified by the European Society of Thoracic Surgeons
Incidence of surgical complications | 3, 6 and 12 months post randomisation
  as classified by the European Society of Thoracic Surgeons
Incidence of Major Post-operative pulmonary complications | Until discharge from hospital post randomisation eg a maximum of 30 days
  as classified by StEP Core Outcome Measures in Perioperative and Anaesthetic Care
Incidence of Major Post-operative pulmonary complications | 3, 6 and 12 months post randomisation
  as classified by StEP Core Outcome Measures in Perioperative and Anaesthetic Care
Incidence of critical care admission | 3, 6 and 12 months post randomisation
  Any admission to critical care extracted from hospital records
Mortality | 3, 6 and 12 months post randomisation
  All deaths due to all causes
Analgesic use | 3, 6 and 12 months post randomisation
  all forms of analgesic use for trial-related pain as reported by patient
Acute pain | Until discharge from hospital post randomisation eg a maximum of 30 days
  Patient reported worst chest pain on visual analogue scale (0-10) with 10 being the worst
Acute pain | Until discharge from hospital post randomisation eg a maximum of 30 days
  Patient reported via Brief Pain Inventory Interference score (0-10, higher = worse)
Acute pain | Until discharge from hospital post randomisation eg a maximum of 30 days
  Patient reported worst chest pain via Short Form McGill Pain Score (0-10 higher = worse score)
Acute pain | 3, 6 and 12 months post randomisation
  Patient reported worst chest pain on visual analogue scale (0-10) with 10 being the worst
Acute pain | 3, 6 and 12 months post randomisation
  Patient reported worst chest pain via Brief Pain Inventory Interference Score (0-10 higher = worse score)
Acute pain | 3, 6 and 12 months post randomisation
  Patient reported worst chest via Short Form McGill Pain Score (0-10 higher = worse score)
Health resource use | Until discharge from hospital post randomisation eg a maximum of 30 days
  Targeted collection of health resource use data from hospital records
Health resource use | 3, 6 and 12 months post randomisation
  Targeted collection of health resource use data from hospital records
General health-related quality of life Index Score | 3, 6 and 12 months post randomisation
  Patient reported using EQ-5D-5L questionnaire Index Score (1.0 = best outcome)
General health-related quality of life Thermometer Score | 3, 6 and 12 months post randomisation
  Patient reported using EQ-5D-5L questionnaire Thermometer Score (0-100, 100 = best outcome)
General health-related quality of life | Until discharge from hospital post randomisation eg a maximum of 30 days
  Patient reported using Hospital Anxiety and Depression Score (0-21, lower = better)
General health-related quality of life | 3, 6 and 12 months post randomisation
  Patient reported using Hospital Anxiety and Depression Score (0-21, lower = better)
Patient Satisfaction with care provided | Until discharge from hospital post randomisation eg a maximum of 30 days
  Patient reported on Likert scale (Very dissatisfied/ Dissatisfied/ Satisfied/ Very satisfied)
Patient Satisfaction with care provided | 3, 6 and 12 months post randomisation
  Patient reported on Likert scale (Very dissatisfied/ Dissatisfied/ Satisfied/ Very satisfied)
Incidence of Serious Adverse Events | 3, and 6 months post randomisation
  Protocol-defined events meeting the accepted trial definition of "serious"

CONTACTS AND LOCATIONS:
Overall Officials: Fang Gao Smith, MD, Principal Investigator — University of Birmingham
Locations (1):
- Heartlands Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The final data set itself will only be available to the direct TOPIC 2 Trial Team, including the Trial Steering Committee (TSC), in the first instance. It will also be made available upon formal request when the reason for the request is approved by the TSC.

REFERENCES:
- [Derived] Shelley B, Goebel A, Grant S, Jackson L, Jarrett H, Jepson M, Kerr A, Marczin N, Mehta R, Melody T, Middleton L, Naidu B, Szentgyorgyi L, Tearne S, Watkins B, Wilson M, Worrall A, Yeung J, Smith FG. Study protocol for a randomised controlled trial to investigate the effectiveness of thoracic epidural and paravertebral blockade in reducing chronic post-thoracotomy pain: 2 (TOPIC 2). Trials. 2023 Nov 23;24(1):748. doi: 10.1186/s13063-023-07463-1. PMID 37996898